CLINICAL TRIAL: NCT00602901
Title: Elderly Back Pain: Comparing Chiropractic to Medical Care
Acronym: HRSA4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18HP01423
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Subacute Low Back Pain; Chronic Low Back Pain
MeSH Terms: interventions — Celecoxib; Naproxen; valdecoxib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- HVLA-SM (Experimental): High-velocity low amplitude spinal manipulation (HVLA-SM)
  Interventions: Other: HVLA-SM
- LVVA-SM (Experimental): Low-velocity variable amplitude spinal manipulation (LVVA-SM)
  Interventions: Other: LVVA-SM
- Usual Medical Care (Active Comparator): Usual medical care - (Celebrex, Aleve, Bextra, Naproxen)
  Interventions: Drug: Usual medical care

INTERVENTIONS:
Other: HVLA-SM — High-velocity low amplitude spinal manipulation (HVLA-SM)
  Arms: HVLA-SM
Other: LVVA-SM — Low-velocity variable amplitude spinal manipulation (LVVA-SM)
  Arms: LVVA-SM
Drug: Usual medical care — Celebrex: po, 200mg, qd, six weeks; Aleve: po, 220mg, bid, six weeks; Bextra: po, 10mg, qd, six weeks; Naproxen: po, 500mg, bid, six weeks.
  Other Names: (Celebrex, Aleve, Bextra, Naproxen)
  Arms: Usual Medical Care

SUMMARY:
The purpose of this study is to compare the clinical effectiveness of two types of chiropractic spinal manipulation to conservative medical care for patients at least 55 years old with sub-acute or chronic low back pain (LBP).

DETAILED DESCRIPTION:
Despite the high prevalence of LBP and the associated economic costs, disability, and lost productivity, and despite the development of several treatment guidelines, one of which recommends chiropractic spinal manipulation for some subgroups of patients with pack pain, the management of LBP remains controversial and highly variable across professions and geographic regions. Although one recent publication describes the design of chiropractic and exercise for seniors with low back or neck pain, no published studies to our knowledge, have assessed the effectiveness of chiropractic manipulation compared to medical care for older adults with sub-acute or chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or older
* Idiopathic low back pain (LBP) of at least four weeks duration
* Meet the diagnostic classification of 1, 2, or 3 according to the Quebec Task Force on Spinal Disorders

Exclusion Criteria:

* Low back pain (LBP) not meeting Quebec Task Force Diagnostic Classifications 1, 2 or 3, especially LBP associated with: frank radiculopathy, altered lower extremity reflex, dermatomal sensory deficit, progressive unilateral muscle weakness or motor loss, symptoms of cauda equina compression, and CT or MRI evidence of anatomical pathology (e.g. abnormal disc, lateral or central stenosis.
* Co-morbid conditions or general poor health that could significantly complicate the prognosis of LBP, including pregnancy, bleeding disorders, extreme obesity, and clear evidence of narcotic or other drug abuse.
* Major clinical depression defined as scores greater that 29 on the Beck Depression Inventory - Second Edition
* Bone or joint pathology that contraindicate spinal manipulative therapy of joint pathology that contraindicate spinal manipulative therapy of the arthropathies and significant osteoporosis
* Pacemaker, because there are safety issues with equipment used to collect data in the biomechanical testing laboratory
* Current or pending litigation related to current episode of LBP.
* Receiving disability for any health-related condition
* Spinal Manipulative care for any reason within the past month
* Unwilling to postpone use of manual therapies for LBP except those provided in the study for the duration of the study period.
* Unable to read or verbally comprehend English.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire(RMDQ). | 6 weeks

SECONDARY OUTCOMES:
Fear Avoidance Beliefs Questionnaire, physical subscale | 6 weeks, 3 months, 6 months
Visual Analogue Scale for Pain | 6 weeks
Postural Sway | 6 weeks
SF-36, v1, Physical Function subscale | 6 weeks
Posteroanterior Spinal Stiffness | 6 weeks
Sit-to-Stand Maneuver | 6 weeks
Spinal Manipulation | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William C Meeker, DC, M.P.H., Principal Investigator — Palmer College of Chiropractic; Maria A Hondras, DC, MPH, Study Director — Palmer College of Chiropractic
Locations (2):
- United States (2):
  - Palmer Center for Chiropractic Research, Davenport, Iowa
  - The University of Iowa, Iowa City, Iowa

REFERENCES:
- [Result] Hondras MA, Long CR, Cao Y, Rowell RM, Meeker WC. A randomized controlled trial comparing 2 types of spinal manipulation and minimal conservative medical care for adults 55 years and older with subacute or chronic low back pain. J Manipulative Physiol Ther. 2009 Jun;32(5):330-43. doi: 10.1016/j.jmpt.2009.04.012. PMID 19539115
- [Result] Hondras MA, Long CR, Haan AG, Spencer LB, Meeker WC. Recruitment and enrollment for the simultaneous conduct of 2 randomized controlled trials for patients with subacute and chronic low back pain at a CAM research center. J Altern Complement Med. 2008 Oct;14(8):983-92. doi: 10.1089/acm.2008.0066. PMID 18990046